CLINICAL TRIAL: NCT04501666
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy and Safety of Nemolizumab (CD14152) in Subjects With Prurigo Nodularis
Brief Title: Study to Assess the Efficacy and Safety of Nemolizumab (CD14152) in Participants With Prurigo Nodularis (PN)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD.06.SPR.202685; 2019-004293-25 (EudraCT Number)
Record Dates: First submitted 2020-07-30; First posted 2020-08-06 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Prurigo Nodularis
Keywords: Prurigo; Neurodermatitis; Pruritus; Skin diseases
MeSH Terms: conditions — Prurigo; Neurodermatitis; Pruritus; Skin Diseases | interventions — nemolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nemolizumab (Experimental): Participants weighing less than (<) 90 kilogram (kg) received two subcutaneous (SC) injections of 30 milligrams (mg) nemolizumab (60 mg loading dose) at baseline then one SC injection once every 4 weeks (Q4W). Participants weighing greater than or equal to (>=) 90 kg received two SC injections of 30 mg nemolizumab (60 mg total) at baseline (no loading dose) and two SC injections Q4W throughout the treatment period of 16 weeks.
  Interventions: Drug: Nemolizumab 30 mg
- Placebo (Placebo Comparator): Participants weighing < 90 kg received two SC injections of matching placebo at baseline, then one SC injection Q4W. Participants weighing >= 90 kg received two SC injections of matching placebo at baseline, then two SC injections Q4W throughout the treatment period of 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nemolizumab 30 mg — Participants received either 30 mg or 60 mg dose of nemolizumab as SC injection.
  Other Names: CD14152
  Arms: Nemolizumab
Drug: Placebo — Participants received matching placebo as SC injection.
  Arms: Placebo

SUMMARY:
The primary objective was to assess the efficacy of nemolizumab (CD14152) compared to placebo in participants greater than or equal to (>=) 18 years of age with prurigo nodularis (PN) after a 16 week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PN for at least 6 months with: Pruriginous nodular lesions on upper limbs, trunk, and/or lower limbs, at least 20 nodules on the entire body with a bilateral distribution and Investigator Global Assessment (IGA) score more than equal to (>=) 3 (based on the IGA scale ranging from 0 to 4, in which 3 was moderate and 4 is severe) at both the screening and baseline visits.
* Severe pruritus was defined as follows on the PP NRS:

  1. At the screening visit (Visit 1): PP NRS score was >= 7.0 for the 24-hour period immediately preceding the screening visit.
  2. At the baseline visit (Visit 2): Mean of the daily intensity of the PP NRS score was >= 7.0 over the previous week.
* Female participants of childbearing potential (that is [i.e,], fertile, following menarche and until becoming post-menopausal unless permanently sterile) must agree to use at least 1 adequate and approved method of contraception throughout the study and for 12 weeks after the last study drug injection.
* Participant was willing and able to comply with all of the time commitments and procedural requirements of the clinical study protocol, including daily diary recordings by the participant using an electronic handheld device provided for this study.

Exclusion Criteria:

* Body weight less than < 30 kg.
* Chronic pruritus resulting from another active condition other than PN, such as but not limited to scabies, lichen simplex chronicus, psoriasis, atopic dermatitis, contact dermatitis, acne, folliculitis, lichen planus, habitual picking/excoriation disorder, sporotrichosis, bullous autoimmune disease, end-stage renal disease, or cholestatic liver disease (example [e.g.] primary biliary cirrhosis) or diabetes mellitus or thyroid disease that is not adequately treated, as per standard of care.
* Unilateral lesions of prurigo (e.g., only one arm affected).
* History of or current confounding skin condition (e.g., Netherton syndrome, cutaneous T-cell lymphoma [mycosis fungoides or Sezary syndrome], chronic actinic dermatitis, dermatitis herpetiformis).
* Participants with a current medical history of chronic obstructive pulmonary disease and/or chronic bronchitis.
* Neuropathic and psychogenic pruritus such as but not limited to notalgia paresthetica, brachioradial pruritus, small fiber neuropathy, skin picking syndrome, or delusional parasitosis.
* Requiring rescue therapy for PN during the screening period or expected to require rescue therapy within 4 weeks following the baseline visit.
* Positive serology results (hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb], hepatitis C (HCV) antibody with positive confirmatory test for HCV (e.g., polymerase chain reaction [PCR]), or human immunodeficiency virus antibody) at the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (95):
- United States (35):
  - Galderma Investigational Site, Birmingham, Alabama
  - Galderma Investigational Site, Los Angeles, California
  - Galderma Investigational Site, Sacramento, California
  - Galderma Investigational Site, San Diego, California
  - Galderma Investigational Site, Santa Monica, California
  - Galderma Investigational Site, Delray Beach, Florida
  - Galderma Investigational Site, Hollywood, Florida
  - Galderma Investigational Site, Largo, Florida
  - Galderma Investigational Site, Miami, Florida
  - Galderma Investigational Site, Pembroke Pines, Florida
  - Galderma Investigational Site, Tampa, Florida
  - Galderma Investigational Site, Columbus, Georgia
  - Galderma Investigational Site, Macon, Georgia
  - Galderma Investigational Site, Chicago, Illinois
  - Galderma Investigational Site, Lake Bluff, Illinois
  - Galderma Investigational Site, Topeka, Kansas
  - Galderma Investigational Site, Baltimore, Maryland
  - Galderma Investigational Site, Ann Arbor, Michigan
  - Galderma Investigational Site, Saint Joseph, Missouri
  - Galderma Investigational Site, St Louis, Missouri
  - Galderma Investigational Site, New York, New York
  - Galderma Investigational Site, High Point, North Carolina
  - Galderma Investigational Site, Raleigh, North Carolina
  - Galderma Investigational Site, Cleveland, Ohio
  - Galderma Investigational Site, Norman, Oklahoma
  - Galderma Investigational Site, Philadelphia, Pennsylvania
  - Galderma Investigational Site, Johnston, Rhode Island
  - Galderma Investigational Site, Providence, Rhode Island
  - Galderma Investigational Site, Knoxville, Tennessee
  - Galderma Investigational Site, Austin, Texas
  - Galderma Investigational Site, Bellaire, Texas
  - Galderma Investigational Site, Laredo, Texas
  - Galderma Investigational Site, Salt Lake City, Utah
  - Galderma Investigational Site, Springville, Utah
  - Galderma Investigational Site, Fairfax, Virginia
- Austria (3):
  - Galderma Investigational Site, Graz
  - Galderma Investigational Site, Linz
  - Galderma Investigational Site, Vienna
- Canada (3):
  - Galderma Investigational Site, Calgary, AL
  - Galderma Investigational Site, London, Ontario
  - Galderma Investigational Site, Saskatoon, Saskatchewan
- Denmark (2):
  - Galderma Investigational Site, Aarhus
  - Galderma Investigational Site, Hellerup
- Germany (22):
  - Galderma Investigational Site, Aachen
  - Galderma Investigational Site, Augsburg
  - Galderma Investigational Site, Bad Bentheim
  - Galderma Investigational Site, Berlin
  - Galderma Investigational Site, Bonn
  - Galderma Investigational Site, Darmstadt
  - Galderma Investigational Site, Dresden
  - Galderma Investigational Site, Düsseldorf
  - Galderma Investigational Site, Eppendorf
  - Galderma Investigational Site, Erlangen
  - Galderma Investigational Site, Göttingen
  - Galderma Investigational Site, Halle
  - Galderma Investigational Site, Hamburg
  - Galderma Investigational Site, Heidelberg
  - Galderma Investigational Site, Kiel
  - Galderma Investigational Site, Lübeck
  - Galderma Investigational Site, Mainz
  - Galderma Investigational Site, Münich
  - Galderma Investigational Site, Münster
  - Galderma Investigational Site, Oldenburg
  - Galderma Investigational Site, Tübingen
  - Galderma Investigational Site, Würzburg
- Hungary (6):
  - Galderma Investigational Site, Budapest
  - Galderma Investigational Site, Gyula
  - Galderma Investigational Site, Kecskemét
  - Galderma Investigational Site, Szeged
  - Galderma Investigational Site, Szolnok
  - Galderma Investigational Site, Zalaegerszeg
- Italy (10):
  - Galderma Investigational Site, Catania
  - Galderma Investigational Site, Chieti
  - Galderma Investigational Site, Genova
  - Galderma Investigational Site, L’Aquila
  - Galderma Investigational Site, Modena
  - Galderma Investigational Site, Napoli
  - Galderma Investigational Site, Parma
  - Galderma Investigational Site, Perugia
  - Galderma Investigational Site, Roma
  - Galderma Investigational Site, Vicenza
- Poland (9):
  - Galderma Investigational Site, Częstochowa
  - Galderma Investigational Site, Gdansk
  - Galderma Investigational Site, Gdynia
  - Galderma Investigational Site, Katowice
  - Galderma Investigational Site, Lodz
  - Galderma Investigational Site, Poznan
  - Galderma Investigational Site, Rzeszów
  - Galderma Investigational Site, Warsaw
  - Galderma Investigational Site, Wroclaw
- Galderma Investigational Site, Solna, Sweden
- United Kingdom (4):
  - Galderma Investigational Site, Dudley
  - Galderma Investigational Site, Glasgow
  - Galderma Investigational Site, London
  - Galderma Investigational Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized data sets from which results presented are derived.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data availability will begin 6 months after approval of the indication by a regulatory body.
  Data availability will end 5 years from publication of the primary study results article.
Access Criteria: Data will be made available to qualified science and medical researchers upon formal request and submission of research proposal detailing planned analyses. Proposals should be directed to clinical.studies@galderma.com

REFERENCES:
- [Result] Kwatra SG, Yosipovitch G, Legat FJ, Reich A, Paul C, Simon D, Naldi L, Lynde C, De Bruin-Weller MS, Nahm WK, Sauder M, Gharib R, Barbarot S, Szepietowski JC, Conrad C, Fleischer A, Laquer VT, Misery L, Serra-Baldrich E, Lapeere H, Ahmad F, Jabbar Lopez ZK, Piketty C, Stander S; OLYMPIA 2 Investigators. Phase 3 Trial of Nemolizumab in Patients with Prurigo Nodularis. N Engl J Med. 2023 Oct 26;389(17):1579-1589. doi: 10.1056/NEJMoa2301333. PMID 37888917
- [Derived] Stander S, Rodriguez DN, Dias-Barbosa C, Filipenko D, Puelles J, Jabbar-Lopez ZK, Piketty C, Wiegmann H, Kwatra SG. Content Validity and Psychometric Validation of an Adapted Version of the Subject Sleep Diary in Prurigo Nodularis. Dermatol Ther (Heidelb). 2025 Jun;15(6):1405-1426. doi: 10.1007/s13555-025-01406-1. Epub 2025 Apr 23. PMID 40266487
- [Derived] Stander S, Yosipovitch G, Legat FJ, Reich A, Paul C, Simon D, Naldi L, Metz M, Tsianakas A, Pink A, Fage S, Micali G, Weisshaar E, Sundaram H, Metelitsa A, Augustin M, Wollenberg A, Homey B, Fargnoli MC, Sofen H, Korman NJ, Skov L, Chen X, Jabbar-Lopez ZK, Piketty C, Kwatra SG; OLYMPIA 1 Investigators. Efficacy and Safety of Nemolizumab in Patients With Moderate to Severe Prurigo Nodularis: The OLYMPIA 1 Randomized Clinical Phase 3 Trial. JAMA Dermatol. 2025 Feb 1;161(2):147-156. doi: 10.1001/jamadermatol.2024.4796. PMID 39602139
- See also: Description Phase 3 Trial of Nemolizumab in Patients with Prurigo Nodularis — http://www.nejm.org/doi/full/10.1056/NEJMoa2301333

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 77 sites in 10 countries.
Pre-assignment Details: A total of 286 participants were randomized to receive either nemolizumab (CD14152) or placebo.
Groups:
- Nemolizumab: Participants weighing less than (<) 90 kilogram (kg) received two subcutaneous (SC) injections of 30 milligrams (mg) nemolizumab (60 mg loading dose) at baseline then one SC injection once for every 4 weeks (Q4W). Participants weighing greater than or equal to (>=) 90 kg received two SC injections of 30 mg nemolizumab (60 mg total) at baseline (no loading dose) and two SC injections Q4W throughout the treatment period of 16 weeks.
  Nemolizumab: Participants received either 30 mg or 60 mg dose of nemolizumab as SC injection.
Period: Overall Study
Arm/Group | Nemolizumab | Placebo
Started | 190 | 96
Treated | 187 | 95
Completed | 166 | 83
Not Completed | 24 | 13
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 12 | 4
Not completed — Subject's request | 10 | 6
Not completed — Protocol Deviation | 2 | 1
Not completed — Other-- site permanently closing | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent-to-treat population (ITT) population which consisted of all randomized participants.
Groups:
- Nemolizumab: Participants weighing <90 kg received two SC injections of 30 mg nemolizumab (60 mg loading dose) at baseline then one SC injection Q4W. Participants weighing >=90 kg received two SC injections of 30 mg nemolizumab (60 mg total) at baseline (no loading dose) and two SC injections Q4W throughout the treatment period of 16 weeks. Nemolizumab: Participants received either 30 mg or 60 mg dose of nemolizumab as SC injection.
- Placebo: Participants weighing <90 kg received two SC injections of matching placebo at baseline, then one SC injection Q4W. Participants weighing >=90 kg received two SC injections of matching placebo at baseline, then two SC injections Q4W throughout the treatment period of 16 weeks. Placebo: Participants received matching placebo as SC injection.
- Total: Total of all reporting groups
Arm/Group | Nemolizumab | Placebo | Total
Number analyzed (Participants) | 190 | 96 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (12.77) | 57.6 (13.36) | 57.5 (12.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 56 | 166
  Male | 80 | 40 | 120
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 184 | 88 | 272
  Unknown or Not Reported | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 10 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 10 | 28
  White | 160 | 81 | 241
  More than one race | 0 | 0 | 0
  Others | 1 | 2 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Europe | 141 | 71 | 212
  North America | 49 | 25 | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Improvement of Greater Than or Equal to (>=) 4 From Baseline in Weekly Average Peak Pruritus Numeric Rating Scale (PP NRS) at Week 16
Description: The Peak Pruritus NRS is a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores were provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome. Weekly values are calculated as the average of 7 consecutive days of data up to the target study day (excluding) and set to missing if less than 4 days of data are available. Analysis window extension was applied to both timepoints, as described in the SAP. If a participant received any rescue therapy, composite variable strategy is applied, the underlying data at/after receipt of rescue therapy is set as worst possible value, and the response is derived from underlying data value. Participants with missing results are considered as non-responders.
Time Frame: Baseline, Week 16
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 190 | 96
Participants | 111 | 16
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; A hierarchical testing procedure was used to control the overall type I error. Testing was then performed sequentially in order the outcome measures were reported and continued when previous outcome measure was statistically significant at two-sided 0.05; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — A 2-sided p-value was derived from Cochran-Mantel-Haenszel (CMH) test using the randomized stratification variables (analysis center and body weight at randomization [< 90 kg, >= 90 kg]). Threshold of significance at 0.05; Strata adjusted percentage difference = 40.1, 95% CI 2-sided [29.4 to 50.8]

2. Primary Outcome: Number of Participants With an Investigator Global Assessment (IGA) Success at Week 16
Description: IGA success is defined as clear (0) or almost clear (1), and a reduction from baseline of greater than or equal to 2 points at week 16. Full scale is scored from 0-4, higher score indicates more severe symptoms. If a participant received any rescue therapy, composite variable strategy is applied, the underlying data at/after receipt of rescue therapy is set as worst possible value, and the response is derived from underlying data value. Participants with missing results are considered as non-responders.
Time Frame: Baseline, Week 16
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 190 | 96
Participants | 50 | 7
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0025, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Strata adjusted percentage difference = 14.6, 95% CI 2-sided [6.7 to 22.6]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Adverse Events of Special Interest (AESIs), and Serious Adverse Events (SAEs)
Description: AE was defined as any untoward medical occurrence in a clinical study participant administered a medicinal product which does not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs occurring after the first administration of the study drug until the last study visit. SAE was any untoward medical occurrence, in the view of either the Investigator or Sponsor, that resulted in death, was life-threatening, resulted in inpatient hospitalisation or prolongation of existing hospitalisation, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was an important medical event. AESI was a noteworthy TEAE for the study drug that was to be monitored closely and reported promptly. Relatedness to study drug was based on Investigator's discretion. Analysis was performed on safety population which included all randomised participants who received at least 1 administration of study drug.
Time Frame: From Baseline up to end of treatment period (24 weeks)
Population: Safety population included all randomized participants who received at least 1 administration of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 187 | 95
Participants
  TEAEs | 134 | 62
  AESIs | 32 | 18
  SAEs | 16 | 10

4. Secondary Outcome: Number of Participants With an Improvement of >= 4 From Baseline in Weekly Average PP NRS at Week 4
Description: The Peak Pruritus NRS is a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores were provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome. Weekly values are calculated as average of 7 consecutive days data up to the target study day (excluding) and set to missing, if less than 4 days data are available. Analysis window extension was applied to baseline, as described in the SAP. If a participant received any rescue therapy, composite variable strategy is applied, the underlying data at/after receipt of rescue therapy is set as worst possible value, and the response is derived from underlying data value. Participants with missing results are considered as non-responders.
Time Frame: Baseline, Week 4
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 190 | 96
Participants | 78 | 6
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — A 2-sided p-value was derived from CMH test using the randomized stratification variables (analysis center and body weight at randomization [< 90 kg, >= 90 kg]). Threshold of significance at 0.05; Strata adjusted percentage difference = 31.7, 95% CI 2-sided [23.0 to 40.4]

5. Secondary Outcome: Number of Participants With PP NRS < 2 at Week 16
Description: The Peak Pruritus NRS is a scale that was used by the participants to report the intensity of their pruritus (itch) during the last 24 hours. For maximum itch intensity: the scores were provided on a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable'. Higher scores indicate worse outcome. Weekly values are calculated as average of 7 consecutive days data up to the target study day (excluding) and set to missing, if less than 4 days data are available. Analysis window extension was applied to week 16, as described in the SAP. If a participant received any rescue therapy, composite variable strategy is applied, the underlying data at/after receipt of rescue therapy is set as worst possible value, and the response is derived from underlying data value. Participants with missing results are considered as non-responders.
Time Frame: Week 16
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 190 | 96
Participants | 65 | 4
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Strata adjusted percentage difference = 30.5, 95% CI 2-sided [22.3 to 38.7]

6. Secondary Outcome: Number of Participants With an Improvement of >=4 From Baseline in Sleep Disturbance Numeric Rating Scale (SD NRS) at Week 16
Description: The SD NRS is a scale to report the degree of participant sleep loss related to PN. The baseline SD NRS was determined based on the average of daily SD NRS (score ranging from 0 to 10) during the 7 days up to the treatment start (including until treatment start time). A minimum of 4 daily scores out of the 7 days up to baseline study day is required for this calculation. On a scale of 0 to 10, with 0 being 'no sleep loss related to the symptoms of my skin disease (prurigo nodularis)' and 10 being 'I did not sleep at all due to the symptoms of prurigo nodularis'. Higher scores indicate worse outcome. Analysis window extension was applied to both timepoints, as described in the SAP. If a participant received any rescue therapy, composite variable strategy is applied, the underlying data at/after receipt of rescue therapy is set as worst possible value, and the response is derived from underlying data value. Participants with missing results are considered as non-responders.
Time Frame: Baseline, Week 16
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 190 | 96
Participants | 95 | 11
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Strata adjusted percentage difference = 38.0, 95% CI 2-sided [27.8 to 48.2]

7. Secondary Outcome: Number of Participants With an Improvement of >=4 From Baseline in SD NRS at Week 4
Description: SD NRS is a scale to be used by the participants to report the degree of their sleep loss related to PN. The baseline SD NRS was determined based on the average of daily SD NRS (score ranging from 0 to10) during the 7 days up to the treatment start (including until treatment start time). A minimum of 4 daily scores out of the 7 days up to baseline study day is required for this calculation. On a scale of 0 to 10, with 0 being 'no sleep loss related to the symptoms of my skin disease (prurigo nodularis)' and 10 being 'I did not sleep at all due to the symptoms of prurigo nodularis'. Higher scores indicate worse outcome. Analysis window extension was applied to baseline, as described in the SAP. If a participant received any rescue therapy, composite variable strategy is applied, the underlying data at/after receipt of rescue therapy is set as worst possible value, and the response is derived from underlying data value. Participants with missing results are considered as non-responde
Time Frame: Baseline, Week 4
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 190 | 96
Participants | 59 | 5
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Strata adjusted percentage difference = 22.7, 95% CI 2-sided [14.7 to 30.7]

8. Secondary Outcome: Number of Participants With PP NRS < 2 at Week 4
Description: as for outcome 4
Time Frame: Week 4
Population: ITT population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Nemolizumab | Placebo
Number analyzed (Participants) | 190 | 96
Participants | 41 | 1
Statistical Analysis 1: Comparison: Nemolizumab vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Strata adjusted percentage difference = 18.7, 95% CI 2-sided [12.3 to 25.0]

ADVERSE EVENTS:
Time Frame: Baseline up to end of treatment period (24 weeks)
Description: Safety population included all randomized participants who received at least 1 administration of study drug.
Arm/Group | Nemolizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/187 | 1/95
Serious Adverse Events (participants affected / at risk) | 16/187 | 10/95
Other Adverse Events (participants affected / at risk) | 61/187 | 38/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nemolizumab (N=187) | Placebo (N=95)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac sarcoidosis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Arachnoid cyst (Nervous system disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 1 (1) | 0 (0)
Campylobacter colitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nemolizumab (N=187) | Placebo (N=95)
Headache (Nervous system disorders) | 13 (16) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 5 (6)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 15 (17) | 18 (21)
Eczema (Skin and subcutaneous tissue disorders) | 10 (10) | 1 (1)
COVID-19 (Infections and infestations) | 14 (14) | 14 (14)
Nasopharyngitis (Infections and infestations) | 11 (12) | 8 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (12) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT04501666/Prot_002.pdf
  • Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT04501666/SAP_003.pdf